CLINICAL TRIAL: NCT02415465
Title: Continuous Adductor Canal Block (CACB) vs. Combined Spinal Epidural (CSE) in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14090501
Record Dates: First submitted 2015-04-06; First posted 2015-04-14 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Arthroplasty
Keywords: Knee; Replacement
MeSH Terms: interventions — Injections, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Combined Spinal Epidural (Active Comparator): Spinal Intraoperative Anesthesia with standard Epidural (0.1% bupivacaine with fentanyl 5 mcg/mL running at 6mL/hr with 1mL q15 bolus) with standard post-operative analgesics.
  Interventions: Procedure: Epidural; Procedure: Spinal
- General+Continuous Adductor Canal Block (Active Comparator): General Intraoperative Anesthesia with standard post-operative Continuous Adductor Canal Block (0.2% ropivacaine running at 6-8mL/hr) with standard post-operative analgesics.
  Interventions: Procedure: Continuous Adductor Canal Block; Procedure: General
- Spinal+Continuous Adductor Canal Block (Active Comparator): Spinal Intraoperative Anesthesia with standard post-operative Continuous Adductor Canal Block (0.2% ropivacaine running at 6-8mL/hr) with standard post-operative analgesics.
  Interventions: Procedure: Continuous Adductor Canal Block; Procedure: Spinal

INTERVENTIONS:
Procedure: Continuous Adductor Canal Block — Continuous Adductor Canal Block (0.2% ropivacaine running at 6-8mL/hr)
  Arms: General+Continuous Adductor Canal Block; Spinal+Continuous Adductor Canal Block
Procedure: General — General Intraoperative Anesthesia
  Arms: General+Continuous Adductor Canal Block
Procedure: Epidural — Epidural (0.1% bupivacaine with fentanyl 5 mcg/mL running at 6mL/hr with 1mL q15 bolus)
  Arms: Combined Spinal Epidural
Procedure: Spinal — Spinal Intraoperative Anesthesia
  Arms: Combined Spinal Epidural; Spinal+Continuous Adductor Canal Block

SUMMARY:
Purpose: Compare continuous adductor canal block (CACB) to Combined Spinal Epidural (CSE) for total knee arthroplasty in terms of mobility, post-operative pain, and analgesic use.

Hypothesis: CACB will provide better mobility than CSE post operatively.

DETAILED DESCRIPTION:
Purpose: Compare continuous adductor canal block (CACB) to Combined Spinal Epidural (CSE) for total knee arthroplasty in terms of mobility, post-operative pain, and analgesic use.

Hypothesis: CACB will provide better mobility than CSE post operatively.

Background/Scientific Review:

Total knee arthroplasty (TKA) is associated with varying degrees of pain post operatively ranging from mild to severe despite the use of comprehensive multimodal analgesic regimens1. Optimizing pain relief is vital for functional recovery after total knee arthroplasty2. Peripheral nerve blocks have been commonly used to improve pain relief and reduce opioid requirements. The addition of nerve blocks involving the femoral nerve have been shown to provide superior pain control3 and shortened hospital stay compared to epidural or intravenous patient controlled analgesia alone1. However, femoral nerve blocks can result in quadriceps weakness leading to functional impairment and an increased risk of falling post operatively4. Unlike Femoral Nerve Blocks (FNB), adductor canal blocks (ACB) are predominantly sensory blocks which preserve quadriceps muscle strength and ambulation ability better than FNBs, while providing equivalent pain relief5-9.

Recent randomized studies have also shown ACB to be superior to placebo in the setting of spinal and general intraoperative anesthesia in terms of ambulation, pain control, and opioid consumption10-12. In a recent retrospective cohort study, the addition of ACB to local infiltration analgesia (LIA) was associated with further improvement in early ambulation benchmarks and a higher rate of home discharge compared with only LIA9. While CACB and CSE are used as part of routine care at Rush University Medical Center and around the country, there have been no studies directly comparing CACB to CSE.

Study Design: Department funded, single center, prospective, randomized, parallel outcome based clinical trial. 300 subjects scheduled to undergo primary unilateral TKA will be randomized to receive CSE, CACB + General, or CACB + Spinal as per routine care. Subjects will be enrolled for no more than 6 weeks.

Power Analysis: Sample size calculations were based on the primary aim, of CACB plus Spinal anesthesia versus standard care (combined spinal epidural, CSE) improving ambulation distance at postoperative day 1 (POD1). Based on results from a pilot study we found that the CSE group had at POD1 a mean distance traveled of 159 feet with a standard deviation (SD) of 111 feet, while the CACB + Spinal anesthesia subjects walked over twice the distance on average with a similar SD.

To be conservative we expect both the CACB + Spinal anesthesia and CACB + General Anesthesia groups to walk at least 35% farther on average, or at least equal to CSE group.

Based on a one-way, 3-level AVOVA with the primary contrast of CABC + Spinal versus CSE at a 35% greater ambulation difference, for 90% power, with α of 5%, requires a sample size of 84 subjects per group. Increasing the sample size to 100 will provide for a 16% dropout rate. Total of 300 patients.

Treatment Groups:

1. General Intraoperative Anesthesia with standard post-operative Continuous Adductor Canal Block (0.2% ropivacaine running at 6-8mL/hr) with standard post-operative analgesics.
2. Spinal Intraoperative Anesthesia with standard post-operative Continuous Adductor Canal Block (0.2% ropivacaine running at 6-8mL/hr) with standard post-operative analgesics.
3. Spinal Intraoperative Anesthesia with standard Epidural (0.1% bupivacaine with fentanyl 5 mcg/mL running at 6mL/hr with 1mL q15 bolus) with standard post-operative analgesics.

Demographics/Patient Specifics: Age, Sex, ASA score, Weight, Height, Operative Time, BMI, Walker, Cane, Unassisted Ambulation

Risks/Benefits:

Combined spinal epidural anesthesia, general anesthesia, and continuous adductor canal blocks are part of routine anesthesia care at Rush University Medical Center and around the country. Post-operative analgesia regiments are standard of care.

Risks of general anesthesia include sore throat, nausea/vomiting, potential tooth damage, vocal cord injury, mental confusion, awareness, stroke, death. Risks of regional anesthesia (spinal) include bleeding (spinal hematoma), infection (meningitis), nerve damage, headache, hypotension, difficulty urinating, and seizures. There is no difference between epidural catheter and adductor canal catheter in terms of risks, other than the adductor canal catheter carries no risk of headache. These risks are present regardless of the study since either general or spinal anesthesia is used in all total knee arthroplasty procedures.

The only risk involved in participating in the study is the potential for breach of confidentiality and/or privacy. Below is a description of the procedure for maintaining confidentiality. There is no direct benefit to the participants in this study.

Procedures for Maintaining Confidentiality A breach of confidentiality and/or privacy is a risk of this study. To prevent this, all collected data will be stored electronically in password-protected files to protect patient identity and information. All information will be collected and reviewed by the research team only. Data will be maintained on a password-protected computer that will be accessible only to the study team. No patient identifiers will be maintained in the database.

ELIGIBILITY:
Inclusion Criteria:

* Any patient scheduled for a primary unilateral TKA.

Exclusion Criteria:

* Partial knee replacement,
* chronic opioid use,
* history of alcohol or drug abuse,
* preexisting neuropathy in operative limb,
* allergy to local anesthetics,
* ASA Class >3,
* patients who decline to participate,
* BMI >40,
* sleep apnea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Ambulation Distance in feet | daily after surgery until discharge from hospital, expected average up to 5 days
  Patient ambulation distance will be measured daily after surgery until discharge from hospital

SECONDARY OUTCOMES:
Straight Leg Raise | daily after surgery until discharge from hospital, expected average up to 5 days
  Patient's ability to perform straight leg raise daily after surgery until discharge from hospital.
Quadriceps strength | daily after surgery until discharge from hospital, expected average up to 5 days
  Quadriceps strength evaluated using a standard non-invasive handheld dynamometer once pre-operatively and daily after surgery until discharged from hospital.
Pain as measured by numeric pain score | daily after surgery until discharge from hospital, expected average up to 5 days
  Post-operative numeric pain scores during rest and with activity during daily inpatient physical therapy sessions until discharge from hospital
Post-operative inpatient opioid consumption (morphine equivalents) | daily after surgery until discharge from hospital, expected average up to 5 days
  Post-operative inpatient opioid consumption (morphine equivalents) measured daily after surgery until discharge from hospital.
Surgery Complications and Adverse Events during inpatient stay | daily after surgery until discahrge from hospital, expected average up to 5 days
  Surgery Complications and Adverse Events during inpatient stay
  1. Respiratory depression
  2. Sedation
  3. Nausea
  4. Emesis
  5. Motor Blockade
  6. Pruritus
  7. Urinary Retention
  8. Hypotension
  9. Numbness
  10. Falls
  11. DVT or PE
  12. Catheter Site Infection
  13. Block Success

CONTACTS AND LOCATIONS:
Overall Officials: Craig J Della Valle, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States